CLINICAL TRIAL: NCT03833050
Title: The TOGETHER Project - Transplant Organ Genomics to Help Prevent Rejection in Heart Transplant Recipients
Brief Title: The TOGETHER Project - Heart
Acronym: TOGETHER
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Naveen L. Pereira, Principal Investigator, Mayo Clinic
Other Study IDs: 17-000682
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Heart Transplant Rejection
Keywords: heart transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 15 ml peripheral Blood samples will be processed for DNA extraction and plasma for RNA seq isolation peripheral blood assay will be obtained at 1, 3, 6, 12 months and for cause.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Transplant Recipients: Heart Transplant Recipients meeting the criteria for enrollment and consented will be followed post transplant for 1 year after enrollment into the study.
  Blood samples will be obtained at their 1, 3, 6, 12 months and any for cause heart biopsy's obtained. There will be no active intervention for recipients that are enrolled. Results from the samples will not be obtained in real time.

SUMMARY:
The researchers are trying to develop a way to measure the risk of transplant rejection with a blood test.

DETAILED DESCRIPTION:
The study will utilize peripheral blood assays collected at time points that are considered standard of care at most institutions. Subjects will have peripheral blood collected at 1 month, 3 months, 6 months, and 12 months after heart transplantation, as well as any for cause time points. These samples will then be used for purposes of developing an RNA-seq based peripheral blood assay in adult heart transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for enrollment as study participants:

* Adult (≥18 years) solitary heart transplant recipient
* Patient is willing and able to provide informed written consent

Exclusion Criteria:

Patients who meet any of these criteria are not eligible for enrollment as study participants:

* Adult (<18 years) heart transplant recipient
* Patient refusal to enroll in the studyc3. Any simultaneous heart and extra organ transplant, including pancreas, liver, lung, kidney, etc. Subjects who have had previous transplants may be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
RNA-seq based peripheral blood assay in heart transplant recipients | 3 years
  Cases will be reviewed and a subset of the peripheral blood specimens will be sent to Mayo Clinic Laboratories for development of the RNA-seq signature. The number of specimens analyzed will be determined based on the incidence of rejection and the incidence of biopsies for cause needed to develop the signature.

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Pereira, M.D., Principal Investigator — Mayo Clinic; Mark D Stegall, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials